CLINICAL TRIAL: NCT04833010
Title: Effects of Face Coverings During Physical Activity
Brief Title: Effects of Face Masks During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Simon Driver, Research Center Director - The STAR at Frisco, Baylor Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 020-353
Record Dates: First submitted 2021-02-09; First posted 2021-04-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Cardiopulmonary; Exercise; Cognitive Performance; Covid19
MeSH Terms: conditions — Motor Activity; COVID-19 | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No cloth face mask (Active Comparator): Cross-over randomization. Participants randomized to this arm will not wear a cloth face mask for Test 1 which they do a progressive step-exercise cycling test to exhaustion
  Interventions: Other: Cardiopulmonary Exercise Test; Other: Cognitive Performance Test
- Cloth face mask (Experimental): Cross-over randomization. Participants randomized to this arm will wear a cloth face mask for Test 1 which they do a progressive step-exercise cycling test to exhaustion
  Interventions: Other: Cardiopulmonary Exercise Test; Other: Cognitive Performance Test

INTERVENTIONS:
Other: Cardiopulmonary Exercise Test — Participants will complete a Cardiopulmonary Exercise test on cycle ergometer in which they will perform progressive step-exercise cycling to exhaustion
Other: Cognitive Performance Test — Cognitive Performance will be tested using a cognition application on an iPad during the Cardiopulmonary Exercise Test.

SUMMARY:
To describe the primary and secondary outcomes of athletes during a Cardiopulmonary Exercise Test (CPET) on a cycle ergometer with and without a face mask.

ELIGIBILITY:
Inclusion Criteria:

* Be able to come to Baylor Scott & White Sports Therapy and Research at The Star in Frisco, Texas twice in three weeks.
* Be willing to wear a face mask during exercise capacity testing on a stationary bicycle.

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
VO2 max during cardiopulmonary exercise testing on a cycle ergometer | Week 1
  Exercise capacity measured by Cosmed K5 metabolic equipment
VO2 max during cardiopulmonary exercise testing on a cycle ergometer | Week 2
  Exercise capacity measured by Cosmed K5 metabolic equipment
Test duration (time) of cardiopulmonary exercise test on a cycle ergometer | Week 1
  Total time of test
Test duration (time) of cardiopulmonary exercise test on a cycle ergometer | Week 2
  Total time of test
Reaction time of cognitive performance testing during cardiopulmonary exercise test on a cycle ergometer | Week 1
  Cognitive testing will take place at the end of each stage of the CPET. Cognitive testing using the SACL Cognition application on iPad will include a baseline SRT measurement and additional measurements at the end of each stage of the CPET. The baseline will include a 30s session of SRT for familiarization and then a 30s session will be scored. SRT will then be administered for 30s at the end of each stage of the CPET. The SRT task includes a visual stimulus presented on the touchscreen. Subjects will be instructed to press the stimulus on-screen as quickly as possible. Reaction time will be measured on the SRT task. Reaction time is calculated as the average amount of time in seconds between stimulus presentation and user response within a session.
Reaction time of cognitive performance testing during cardiopulmonary exercise test on a cycle ergometer | Week 2
  Cognitive testing will take place at the end of each stage of the CPET. Cognitive testing using the SACL Cognition application on iPad will include a baseline SRT measurement and additional measurements at the end of each stage of the CPET. The baseline will include a 30s session of SRT for familiarization and then a 30s session will be scored. SRT will then be administered for 30s at the end of each stage of the CPET. The SRT task includes a visual stimulus presented on the touchscreen. Subjects will be instructed to press the stimulus on-screen as quickly as possible. Reaction time will be measured on the SRT task. Reaction time is calculated as the average amount of time in seconds between stimulus presentation and user response within a session.
Accuracy of cognitive performance testing during cardiopulmonary exercise test on a cycle ergometer | Week 1
  Cognitive testing will take place at the end of each stage of the CPET. Cognitive testing using the SACL Cognition application on iPad will include a baseline SRT measurement and additional measurements at the end of each stage of the CPET. The baseline will include a 30s session of SRT for familiarization and then a 30s session will be scored. SRT will then be administered for 30s at the end of each stage of the CPET. The SRT task includes a visual stimulus presented on the touchscreen. Subjects will be instructed to press the stimulus on-screen as quickly as possible. Accuracy will be measured on the SRT task. Accuracy is calculated as the total number of correct responses to stimuli divided by the total number of stimuli presented during a session (presented as a percentage).
Accuracy of cognitive performance testing during cardiopulmonary exercise test on a cycle ergometer | Week 2
  Cognitive testing will take place at the end of each stage of the CPET. Cognitive testing using the SACL Cognition application on iPad will include a baseline SRT measurement and additional measurements at the end of each stage of the CPET. The baseline will include a 30s session of SRT for familiarization and then a 30s session will be scored. SRT will then be administered for 30s at the end of each stage of the CPET. The SRT task includes a visual stimulus presented on the touchscreen. Subjects will be instructed to press the stimulus on-screen as quickly as possible. Accuracy will be measured on the SRT task. Accuracy is calculated as the total number of correct responses to stimuli divided by the total number of stimuli presented during a session (presented as a percentage).

SECONDARY OUTCOMES:
Subjective dyspnea rating during cardiopulmonary exercise testing on a cycle ergometer | Week 1
  The Modified Borg Dyspnea Scale (0-10) will be used to assess subjective shortness of breath. Measured during each stage of the exercise protocol during cardiopulmonary exercise test on a cycle ergometer.
Subjective dyspnea rating during cardiopulmonary exercise testing on a cycle ergometer | Week 2
  The Modified Borg Dyspnea Scale (0-10) will be used to assess subjective shortness of breath. Measured during each stage of the exercise protocol during cardiopulmonary exercise test on a cycle ergometer.
Ratings of perceived exertion during cardiopulmonary exercise testing on a cycle ergometer | Week 1
  The Borg Rating of Perceived Exertion (6-20) scale will be used during the test to assess subjective exertion. Measured during each stage of the exercise protocol during cardiopulmonary exercise test on a cycle ergometer
Ratings of perceived exertion during cardiopulmonary exercise testing on a cycle ergometer | Week 2
  The Borg Rating of Perceived Exertion (6-20) scale will be used during the test to assess subjective exertion. Measured during each stage of the exercise protocol during cardiopulmonary exercise test on a cycle ergometer
Oxygen saturation during cardiopulmonary exercise testing on a cycle ergometer | Week 1
  Measured by a pulse oximeter during each stage of the exercise protocol of the cardiopulmonary exercise test on a cycle ergometer
Oxygen saturation during cardiopulmonary exercise testing on a cycle ergometer | Week 2
  Measured by a pulse oximeter during each stage of the exercise protocol of the cardiopulmonary exercise test on a cycle ergometer
Blood lactate during cardiopulmonary exercise testing on a cycle ergometer | Week 1
  Blood lactate will be measured pre and post-CPET using a Nova Medical Lactate Plus: Blood Lactate Measuring Meter-Version 2 device.
Blood lactate during cardiopulmonary exercise testing on a cycle ergometer | Week 2
  Blood lactate will be measured pre and post-CPET using a Nova Medical Lactate Plus: Blood Lactate Measuring Meter-Version 2 device.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Sports Therapy & Research at The Star, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Considered upon request.

REFERENCES:
- See also: Baylor Scott & White Sports Therapy and Research at The Star — https://www.bswhealth.com/Star

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT04833010/Prot_SAP_000.pdf